CLINICAL TRIAL: NCT04436744
Title: A Randomized, Multicenter, Open-Label, Two-Arm, Phase II, Neoadjuvant Study Evaluating the Efficacy, Safety, and Pharmacokinetics of GDC-9545 Plus Palbociclib Compared With Anastrozole Plus Palbociclib for Postmenopausal Women With Estrogen Receptor-Positive and HER2-Negative Untreated Early Breast Cancer
Brief Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Giredestrant Plus Palbociclib Compared With Anastrozole Plus Palbociclib for Postmenopausal Women With Estrogen Receptor-Positive and HER2-Negative Untreated Early Breast Cancer (coopERA Breast Cancer)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO42133; 2020-001007-16 (EudraCT Number)
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Results first posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — giredestrant; Anastrozole; palbociclib; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Giredestrant + Palbociclib (Experimental)
  Interventions: Drug: Giredestrant; Drug: Palbociclib; Procedure: Surgery
- Anastrozole + Palbociclib (Active Comparator)
  Interventions: Drug: Anastrozole; Drug: Palbociclib; Procedure: Surgery

INTERVENTIONS:
Drug: Giredestrant — During the window-of-opportunity phase (first 2 weeks) giredestrant will be taken orally once per day (QD) as a single agent. During the neoadjuvant treatment phase, giredestrant will be taken orally QD on Days 1-28 of each 28-day cycle for a total of 4 cycles, in combination with palbociclib.
  Other Names: GDC-9545; RO7197597; RG6171
  Arms: Giredestrant + Palbociclib
Drug: Anastrozole — During the window-of-opportunity phase (first 2 weeks), anastrozole 1 mg will be taken orally QD as a single agent. During the neoadjuvant treatment phase, anastrozole 1 mg will be taken orally QD on Days 1-28 of each 28-day cycle for a total of 4 cycles, in combination with palbociclib.
  Arms: Anastrozole + Palbociclib
Drug: Palbociclib — During the neoadjuvant treatment phase, palbociclib 125 mg will be taken orally QD on Days 1-21 of a 28-day cycle for a total of 4 cycles.
Procedure: Surgery — Surgery must be performed within a maximum of 14 days after the final cycle in the neoadjuvant treatment phase and ideally should occur as soon as possible after the last dose of study treatment.

SUMMARY:
This is a randomized, multicenter, open-label, two-arm, Phase II study to evaluate the efficacy, safety, and pharmacokinetics of giredestrant versus anastrozole (in the window-of-opportunity phase) and giredestrant plus palbociclib compared with anastrozole plus palbociclib (in the neoadjuvant phase) in postmenopausal women with untreated, estrogen receptor (ER)-positive, human epidermal growth factor receptor-2 (HER2)-negative, early breast cancer.

The study consists of a screening period of up to 28 days, a window-of-opportunity phase for 14 days, followed by a neoadjuvant treatment phase for 16 weeks (four 28-day cycles), surgery, and an end of study visit (28 days after the final dose of study treatment).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women age ≥18 years
* Histologically confirmed operable or inoperable invasive breast carcinoma
* Candidate for neoadjuvant treatment and considered appropriate for endocrine therapy
* Willingness to undergo breast surgery after neoadjuvant treatment and to provide three mandatory tumor samples
* Documented estrogen receptor (ER)-positive tumor in accordance to American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines (Allison et al.2020), assessed locally and defined as ≥1% of tumor cells stained positive on the basis of the most recent tumor biopsy
* Documented progesterone receptor status (positive or negative) as per local assessment
* Documented human epidermal growth factor receptor-2 (HER2)-negative tumor in accordance to 2018 ASCO/CAP guidelines (Wolff et al. 2018), assessed locally on the most recent tumor biopsy
* Ki67 score ≥5% analyzed centrally or locally
* Eastern Cooperative Oncology Group Performance Status 0-1
* Adequate organ function

Exclusion Criteria:

* Stage IV (metastatic) breast cancer
* Inflammatory breast cancer (cT4d)
* Bilateral invasive breast cancer
* History of invasive breast cancer, ductal carcinoma in situ or lobular carcinoma in situ and other malignancy within 5 years prior to screening
* Previous systemic or local treatment for the primary breast cancer currently under investigation
* History of any prior treatment with aromatase inhibitors (AIs), tamoxifen, selective estrogen receptor down regulator, or cyclin-dependent kinase 4 and 6 inhibitors
* Major surgery within 4 weeks prior to randomization
* Known clinically significant history of liver disease consistent with Child-Pugh Class B or C, including hepatitis
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
* History of allergy to anastrozole, or palbociclib or any of its excipients
* Known issues with swallowing oral medication
* History of documented hemorrhagic diathesis, coagulopathy, or thromboembolism
* Active cardiac disease or history of cardiac dysfunction
* Current treatment with medications that are well known to prolong the QT interval
* Active inflammatory bowel disease or chronic diarrhea, short bowel syndrome, or major upper gastrointestinal surgery including gastric resection
* Treatment with strong CYP3A4 inhibitors or inducers within 14 days or 5 drug elimination half-lives prior to randomization
* Known HIV infection
* Serious infection requiring oral or IV antibiotics, or other clinically significant infection within 14 days prior to screening
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (65):
- United States (10):
  - UCLA - Burbank, Burbank, California
  - UCLA - Laguna Hills, Laguna Hills, California
  - UCLA Hematology/Oncology-San Luis Obispo, San Luis Obispo, California
  - UCLA Hematology Oncology-Santa Monica, Santa Monica, California
  - Torrance Memorial Physician Network/Cancer Care, Torrance, California
  - Orlando Health Inc., Orlando, Florida
  - SCRI Florida Cancer Specialists East, West Palm Beach, Florida
  - Saint Barnabas Medical Center Cancer Center, Livingston, New Jersey
  - Tennessee Oncology; Sarah Cannon Research Institute, Nashville, Tennessee
  - Univ of Wisconsin-Madison; Clinical Science Center, Madison, Wisconsin
- Australia (2):
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Westmead Hospital; Medical Oncology and Pallative Care, Westmead, New South Wales
- Brazil (4):
  - Hospital do Cancer de Pernambuco - HCP, Recife, Pernambuco
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Clinica de Pesquisa e Centro de Estudos em Oncologia Ginecologica e Mamaria Ltda, São Paulo, São Paulo
  - Núcleo de Pesquisa São Camilo; ONCOLOGIA CLINICA / QUIMIOTERAPIA, São Paulo, São Paulo
- Germany (3):
  - Universitätsklinikum Dresden, Dresden
  - LUISENKRANKENHAUS; Senological Oncology, Düsseldorf
  - UNIVERSITATSKLINIKUM ERLANGEN; Department of Gynecology and Obstetrics, Erlangen
- Hungary (2):
  - Bacs-Kiskun Megyei Korhaz, SZTE AOK Oktato Korhaza, Onkoradiologiai Kozpont; Onkoradiologiai Kozpont, Kecskemét
  - Tolna Megyei Kórház, Onkológia, Szekszárd
- Poland (4):
  - Szpital Morski Im. Pck; Oncology & Radiotherapy Dept, Gdynia
  - COZL Oddzial Onkologii Klinicznej z pododdzialem Chemioterapii Dziennej, Lublin
  - Centrum Onkologii - Inst.Im. Marii Sklodowskiej-Curie; Oncology, Warsaw
  - DOLNOSLASKIE CENTRUM ONKOLOGII; Oddzial Chirurgii Piersi, Wroclaw
- Russia (6):
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - Private Healthcare Institution Clinical Hospital RZhD Medicine, Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary of Ministry of Healthcare of Tatarstan Republic, Kazan', Tatarstan Republic
  - Filial #1 Regional Oncology Dispensary of Nizhniy Novgorod, Nizhny Novgorod
  - FSI "SRC of Oncology n. a. N.N.Petrov of Rosmedtekhnologiy", Saint Petersburg
  - S-Pb clinical scientific practical center of specialized kinds of medical care (oncological), Saint Petersburg
- South Korea (6):
  - National Cancer Center; Medical Oncology, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Severance Hospital; Internal Medicine, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
- Spain (20):
  - Institutio Catalan De Oncologia, Badalona, Barcelona
  - Complejo Hospitalario de Althaia; Servicio de Oncologia, Manresa, Barcelona
  - Hospital de Jerez de la Frontera; Servicio de Oncologia, Jerez de la Frontera, Cadiz
  - Hospital Universitari Arnau de Vilanova, Lleida, Lerida
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital de Navarra; Servicio de Oncologia, Navarra, Navarre
  - Hospital Universitari Sant Joan de Reus; Planta baja, color lila, Reus, Tarragona
  - Hospital Universitario de Canarias;servicio de Oncologia, San Cristóbal de La Laguna, Tenerife
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Quirón Dexeus, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen de las Nieves : Hospital General, Granada
  - Hospital Clinico San Cecilio, Granada
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario La Paz, Madrid
  - Fundación Jimenez Díaz, Madrid
  - Hosp Univ Fundacion Alcorcon, Madrid
  - Hospital Universitario Virgen de La Arrixaca, Murcia
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital General Universitario de Valencia, Valencia
- Taiwan (2):
  - National Cheng Kung Uni Hospital; Surgery, Tainan
  - National Taiwan Uni Hospital; General Surgery, Taipei
- Ukraine (6):
  - Regional Oncology Center of Kharkiv Regional Council; Department of Soft Tissues and Breast Cancer, Kharkiv, Kharkiv Governorate
  - Odesa Regional Clinical Hospital; Department of Thoracic Surgery, Odesa, Kharkiv Governorate
  - Khmelnytsky Regional Antitumor Center; Department of Breast, Skin, Soft Tissues and Bones Tumors, Khmelnytskyi, Podolia Governorate
  - Municipal institution Dnipropetrovsk City Multifield Clinical Hospital #4; dept. of Chemotherapy, Dnipropetrovsk
  - ME Kryviy Rih Oncology Dispensary of Dnipropetrovs'k Regional Council; Chemotherapy Department, Kryvyi Rih
  - Kyiv Regional Oncological Dispensary, Kyiv

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Hurvitz SA, Bardia A, Quiroga V, Park YH, Blancas I, Alonso-Romero JL, Vasiliev A, Adamchuk H, Salgado M, Yardley DA, Berzoy O, Zamora-Aunon P, Chan D, Spera G, Xue C, Ferreira E, Badovinac Crnjevic T, Perez-Moreno PD, Lopez-Valverde V, Steinseifer J, Fernando TM, Moore HM, Fasching PA; coopERA Breast Cancer study group. Neoadjuvant palbociclib plus either giredestrant or anastrozole in oestrogen receptor-positive, HER2-negative, early breast cancer (coopERA Breast Cancer): an open-label, randomised, controlled, phase 2 study. Lancet Oncol. 2023 Sep;24(9):1029-1041. doi: 10.1016/S1470-2045(23)00268-1. PMID 37657462

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at 64 investigative sites in Australia, Brazil, Germany, Hungary, Korea, Poland, Russia, Spain, Taiwan, the United States, and Ukraine, from 4 September 2020 to 24 November 2021.
Pre-assignment Details: A total of 264 participants were screened.
Groups:
- Giredestrant + Palbociclib: Participants received giredestrant, 30 milligrams (mg), orally, once per day (QD), during the window-of-opportunity phase of two weeks. During the neoadjuvant treatment phase, participants received giredestrant, 30 mg, orally, QD on Days 1-28 of each 28-day cycle for a total of 4 cycles in combination with palbociclib, 125 mg, administered orally, QD on Days 1-21 of each 28-day cycle for a total of 4 cycles.
- Anastrozole + Palbociclib: Participants received anastrozole, 1 mg, orally, QD, during the window-of-opportunity phase of two weeks. During the neoadjuvant treatment phase, participants received anastrozole, 1 mg, orally, QD on Days 1-28 of each 28-day cycle for a total of 4 cycles in combination with palbociclib, 125 mg, administered orally, QD on Days 1-21 of each 28-day cycle for a total of 4 cycles.
Period: Overall Study
Arm/Group | Giredestrant + Palbociclib | Anastrozole + Palbociclib
Started | 112 | 109
Completed | 108 | 98
Not Completed | 4 | 11
Not completed — Adverse Event | 1 | 1
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Progressive Disease | 0 | 4
Not completed — Protocol Deviation | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all randomized participants.
Groups:
- Giredestrant + Palbociclib: Participants received giredestrant, 30 mg, orally, QD, during the window-of-opportunity phase of two weeks. During the neoadjuvant treatment phase, participants received giredestrant, 30 mg, orally, QD on Days 1-28 of each 28-day cycle for a total of 4 cycles in combination with palbociclib, 125 mg, administered orally, QD on Days 1-21 of each 28-day cycle for a total of 4 cycles.
- Total: Total of all reporting groups
Arm/Group | Giredestrant + Palbociclib | Anastrozole + Palbociclib | Total
Number analyzed (Participants) | 112 | 109 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (7.9) | 62.4 (9.3) | 62.8 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 109 | 221
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 11 | 27
  Not Hispanic or Latino | 95 | 98 | 193
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 9 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 100 | 94 | 194
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9
Ki67 Scores [Mean (Full Range); unit: percent Ki67 score] — Ki67 is a proliferation biomarker with prognostic value in estrogen receptor (ER)-positive breast cancer. Ki67 scores were centrally assessed with immunohistochemistry and defined as a percentage of positively stained tumor cell nuclei among the total number of tumor cells assessed, with a potential range of 0-100%. A score of 0% indicates no tumor cell nuclei with Ki67 staining and a score of 100% indicates all tumor cell nuclei are positively stained with Ki67. The higher percentage score indicates higher risk of recurrence.
  percent Ki67 score | 37.92 [6.6 to 96.3] | 41.66 [7.8 to 98.9] | 39.76 [6.6 to 98.9]

OUTCOME MEASURES:

1. Primary Outcome: Relative Percent Change in Ki67 Scores From Baseline to Week 2
Description: Ki67 is a proliferation biomarker with prognostic value in ER-positive breast cancer. Ki67 scores were centrally assessed with immunohistochemistry and defined as a percentage of positively stained tumor cell nuclei among the total number of tumor cells assessed, with a potential range of 0-100%. A score of 0% indicates no tumor cell nuclei with Ki67 staining and a score of 100% indicates all tumor cell nuclei are positively stained with Ki67. The relative percentage change was calculated using Ki67 scores at Baseline and Week 2. Relative Percent Change was defined as Week 2 Ki67 percentage score/Baseline Ki67 percentage score*100. A smaller value of relative percentage change indicates improvement.
Time Frame: Baseline, Week 2
Population: Efficacy-evaluable population included participants with Ki67-evaluable tumor specimens at baseline and Week 2. Participants with missing central Ki67 scores at baseline and/or Week 2 were excluded from the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Giredestrant + Palbociclib | Anastrozole + Palbociclib
Number analyzed (Participants) | 107 | 94
percent change | 25 [20 to 30] | 33 [27 to 41]
Statistical Analysis 1: Comparison: Giredestrant + Palbociclib vs Anastrozole + Palbociclib; Test type: Superiority; p = 0.0433, t-test, 2 sided

2. Secondary Outcome: Overall Response Rate (ORR) by Ultrasound as Determined by the Investigator
Description: ORR was defined as the percentage of participants with a complete response (CR) or partial response (PR), as determined by the investigator according to Modified Response Evaluation Criteria in Solid Tumors (mRECIST). Ultrasound and clinical exam were used to assess response. CR per mRECIST was defined as the disappearance of all target lesions. PR per mRECIST was defined as at least 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. An estimate of ORR and its 95% confidence interval (CI) was calculated using the Clopper-Pearson method.
Time Frame: Baseline up to Cycle 4 Day 1 (each cycle is 28 days)
Population: ORR-evaluable population included all randomized participants with measurable disease at baseline. Participants not meeting the criteria for ORR, including participants without any post-baseline tumor assessment, were considered as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Giredestrant + Palbociclib | Anastrozole + Palbociclib
Number analyzed (Participants) | 112 | 108
percentage of participants | 50.0 [40.40 to 59.60] | 49.1 [39.33 to 58.87]
Statistical Analysis 1: Comparison: Giredestrant + Palbociclib vs Anastrozole + Palbociclib; ORR was calculated using the stratified Cochran-Mantel-Haenszel test; Test type: Superiority; p = 0.8272, Cochran-Mantel-Haenszel; Difference in Overall Response Rates = -0.93, 95% CI 2-sided [-14.66 to 12.81]

3. Secondary Outcome: Complete Cell Cycle Arrest (CCCA) Rate at Week 2
Description: CCCA was defined as the percentage of participants with centrally assessed Ki67 scores ≤2.7%. The CCCA rate at Week 2 was summarized.
Time Frame: Week 2
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Giredestrant + Palbociclib | Anastrozole + Palbociclib
Number analyzed (Participants) | 107 | 94
percentage of participants | 19.6 | 12.8
Statistical Analysis 1: Comparison: Giredestrant + Palbociclib vs Anastrozole + Palbociclib; Test type: Superiority; Difference in Rate = 6.86, 95% CI 2-sided [-4.25 to 17.97]

4. Secondary Outcome: Number of Participants With Adverse Events (AEs) With Severity Determined in Accordance With National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)
Description: AE is any untoward medical occurrence in clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable & unintended sign, symptom/disease temporally associated with use of a medicinal product, whether or not related to medicinal product. Preexisting conditions which worsen during a study also considered as AEs. Severity of AEs was determined per NCI CTCAE v5.0. Grade 1: Mild; asymptomatic/mild symptoms; clinical/diagnostic observations only; or intervention not indicated; Grade 2: Moderate; minimal, local/non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living; Grade 3: Severe/medically significant, but not immediately life-threatening: hospitalization/prolongation of hospitalization indicated; disabling/limiting self-care activities of daily living; Grade 4: Life-threatening consequences/urgent intervention indicated; Grade 5: Death related to AE.
Time Frame: From baseline up to 28 days after the last dose (up to approximately 24 weeks)
Population: Safety-evaluable population included all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Giredestrant + Palbociclib | Anastrozole + Palbociclib
Number analyzed (Participants) | 112 | 109
Participants
  AEs | 104 | 98
  Grade 1 | 19 | 20
  Grade 2 | 35 | 31
  Grade 3 | 45 | 45
  Grade 4 | 4 | 2
  Grade 5 | 1 | 0

5. Secondary Outcome: Change From Baseline in Respiratory Rate Over Time
Description: Respiratory rate was measured while the participant was in a seated position.
Time Frame: Baseline; Cycles 1-2: Day 1 and Day 15; Cycles 3-4: Day 1; day of surgery (up to 2 weeks after the final dose of study treatment [approximately Week 18]) and end of study (up to approximately 24 weeks)
Population: Safety-evaluable population included all participants who received any amount of study treatment. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: breath/minute (min)
Groups:
- Giredestrant + Palbociclib: Participants received giredestrant 30 mg, orally, QD, during the window-of-opportunity phase of two weeks. During the neoadjuvant treatment phase, participants received giredestrant, 30 mg, orally, QD on Days 1-28 of each 28-day cycle for a total of 4 cycles in combination with palbociclib, 125 mg, administered orally, QD on Days 1-21 of each 28-day cycle for a total of 4 cycles.
Arm/Group | Giredestrant + Palbociclib | Anastrozole + Palbociclib
Number analyzed (Participants) | 98 | 102
breath/minute (min)
  Baseline | 17.16 (2.27) | 17.10 (2.05)
  Change from Baseline at Cycle 1 Day 1: number analyzed (Participants) | 91 | 91
  Change from Baseline at Cycle 1 Day 1 | 0.30 (2.12) | 0.26 (1.50)
  Change from Baseline at Cycle 1 Day 15: number analyzed (Participants) | 90 | 88
  Change from Baseline at Cycle 1 Day 15 | -0.01 (1.49) | -0.06 (1.36)
  Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 89 | 92
  Change from Baseline at Cycle 2 Day 1 | -0.10 (1.83) | 0.16 (1.34)
  Change from Baseline at Cycle 2 Day 15: number analyzed (Participants) | 89 | 91
  Change from Baseline at Cycle 2 Day 15 | -0.24 (1.71) | -0.03 (1.64)
  Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 87 | 89
  Change from Baseline at Cycle 3 Day 1 | 0.07 (1.58) | 0.01 (1.61)
  Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 91 | 83
  Change from Baseline at Cycle 4 Day 1 | -0.04 (1.71) | 0.01 (1.53)
  Change from Baseline at Day of Surgery: number analyzed (Participants) | 72 | 62
  Change from Baseline at Day of Surgery | 0.04 (1.72) | -0.02 (1.69)
  Change from Baseline at End of Study: number analyzed (Participants) | 88 | 81
  Change from Baseline at End of Study | -0.26 (1.65) | 0.01 (1.42)

6. Secondary Outcome: Change From Baseline in Pulse Rate Over Time
Description: Pulse rate was measured while the participant was in a seated position.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Giredestrant + Palbociclib | Anastrozole + Palbociclib
Number analyzed (Participants) | 98 | 102
beats/min
  Baseline | 75.86 (10.67) | 76.73 (9.85)
  Change from Baseline at Cycle 1 Day 1: number analyzed (Participants) | 90 | 92
  Change from Baseline at Cycle 1 Day 1 | -4.74 (9.07) | -1.96 (9.43)
  Change from Baseline at Cycle 1 Day 15: number analyzed (Participants) | 91 | 90
  Change from Baseline at Cycle 1 Day 15 | -6.02 (12.02) | -1.47 (8.15)
  Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 90 | 92
  Change from Baseline at Cycle 2 Day 1 | -5.20 (10.26) | -1.11 (10.79)
  Change from Baseline at Cycle 2 Day 15: number analyzed (Participants) | 92 | 91
  Change from Baseline at Cycle 2 Day 15 | -7.68 (11.03) | -1.95 (8.64)
  Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 88 | 90
  Change from Baseline at Cycle 3 Day 1 | -5.47 (11.61) | -0.81 (10.83)
  Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 91 | 83
  Change from Baseline at Cycle 4 Day 1 | -5.67 (9.79) | -1.11 (10.62)
  Change from Baseline at Day of Surgery: number analyzed (Participants) | 73 | 65
  Change from Baseline at Day of Surgery | -4.14 (11.25) | -1.26 (10.46)
  Change from Baseline at End of Study: number analyzed (Participants) | 88 | 81
  Change from Baseline at End of Study | -0.61 (10.74) | 1.59 (10.44)

7. Secondary Outcome: Change From Baseline in Systolic Blood Pressure Over Time
Description: Systolic blood pressure was measured while the participant was in a seated position.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Giredestrant + Palbociclib | Anastrozole + Palbociclib
Number analyzed (Participants) | 98 | 102
millimeters of mercury (mmHg)
  Baseline | 135.63 (14.13) | 130.03 (16.43)
  Change from Baseline at Cycle 1 Day 1: number analyzed (Participants) | 91 | 92
  Change from Baseline at Cycle 1 Day 1 | -0.82 (11.11) | 1.12 (13.65)
  Change from Baseline at Cycle 1 Day 15: number analyzed (Participants) | 91 | 90
  Change from Baseline at Cycle 1 Day 15 | -2.55 (14.01) | 0.23 (15.85)
  Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 90 | 92
  Change from Baseline at Cycle 2 Day 1 | -2.08 (14.13) | 0.28 (14.43)
  Change from Baseline at Cycle 2 Day 15: number analyzed (Participants) | 92 | 90
  Change from Baseline at Cycle 2 Day 15 | -4.25 (15.37) | 0.16 (16.49)
  Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 88 | 90
  Change from Baseline at Cycle 3 Day 1 | -2.66 (16.95) | 0.33 (15.81)
  Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 91 | 83
  Change from Baseline at Cycle 4 Day 1 | -1.29 (15.30) | -0.25 (14.17)
  Change from Baseline at Day of Surgery: number analyzed (Participants) | 74 | 65
  Change from Baseline at Day of Surgery | -2.35 (13.79) | 1.51 (15.24)
  Change from Baseline at End of Study: number analyzed (Participants) | 88 | 81
  Change from Baseline at End of Study | -5.38 (13.98) | -1.67 (16.20)

8. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure Over Time
Description: Diastolic blood pressure was measured while the participant was in a seated position.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Giredestrant + Palbociclib | Anastrozole + Palbociclib
Number analyzed (Participants) | 98 | 102
mmHg
  Baseline | 80.40 (8.84) | 78.49 (9.55)
  Change from Baseline at Cycle 1 Day 1: number analyzed (Participants) | 91 | 92
  Change from Baseline at Cycle 1 Day 1 | -2.42 (7.77) | 0.39 (8.13)
  Change from Baseline at Cycle 1 Day 15: number analyzed (Participants) | 91 | 90
  Change from Baseline at Cycle 1 Day 15 | -4.80 (8.58) | -2.42 (8.71)
  Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 90 | 92
  Change from Baseline at Cycle 2 Day 1 | -4.79 (10.08) | -0.76 (8.80)
  Change from Baseline at Cycle 2 Day 15: number analyzed (Participants) | 92 | 90
  Change from Baseline at Cycle 2 Day 15 | -5.64 (9.24) | -1.32 (9.64)
  Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 88 | 90
  Change from Baseline at Cycle 3 Day 1 | -5.25 (8.51) | -0.16 (9.52)
  Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 91 | 83
  Change from Baseline at Cycle 4 Day 1 | -4.35 (9.31) | -2.57 (9.50)
  Change from Baseline at Day of Surgery: number analyzed (Participants) | 74 | 65
  Change from Baseline at Day of Surgery | -4.93 (8.72) | -2.15 (9.58)
  Change from Baseline at End of Study: number analyzed (Participants) | 88 | 81
  Change from Baseline at End of Study | -2.73 (8.37) | -2.52 (12.11)

9. Secondary Outcome: Change From Baseline in Body Temperature Over Time
Time Frame: as for outcome 5
Population: Safety-evaluable population included all participants who received any amount of study treatment. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: Celsius (C)
Arm/Group | Giredestrant + Palbociclib | Anastrozole + Palbociclib
Number analyzed (Participants) | 112 | 109
Celsius (C)
  Baseline | 36.35 (0.41) | 36.45 (0.38)
  Change from Baseline at Cycle 1 Day 1: number analyzed (Participants) | 110 | 105
  Change from Baseline at Cycle 1 Day 1 | 0.07 (0.39) | 0.04 (0.36)
  Change from Baseline at Cycle 1 Day 15: number analyzed (Participants) | 107 | 103
  Change from Baseline at Cycle 1 Day 15 | 0.01 (0.41) | -0.01 (0.43)
  Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 108 | 105
  Change from Baseline at Cycle 2 Day 1 | 0.03 (0.40) | -0.04 (0.52)
  Change from Baseline at Cycle 2 Day 15: number analyzed (Participants) | 110 | 102
  Change from Baseline at Cycle 2 Day 15 | -0.03 (0.37) | -0.12 (0.47)
  Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 109 | 102
  Change from Baseline at Cycle 3 Day 1 | -0.04 (0.42) | 0.01 (0.39)
  Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 109 | 103
  Change from Baseline at Cycle 4 Day 1 | -0.03 (0.37) | -0.08 (0.38)
  Change from Baseline at Day of Surgery: number analyzed (Participants) | 97 | 85
  Change from Baseline at Day of Surgery | 0.06 (0.39) | -0.01 (0.38)
  Change from Baseline at End of Study: number analyzed (Participants) | 107 | 102
  Change from Baseline at End of Study | 0.05 (0.39) | -0.04 (0.48)

10. Secondary Outcome: Number of Participants With Shifts in Hematology Test Parameters From NCI-CTCAE Grade 0-2 at Baseline to Grade 3-4 at Post-baseline
Description: Hematology test parameters were measured per NCI CTCAE v5.0. Grade 0 is normal, and Grades 1 to 4 represent worsening levels of the parameter outside of the normal range in the specified direction of the abnormality (high and low are above and below the range, respectively). Number of participants with shift in the hematology values from grade 0-2 at baseline to grade 3-4 at post-baseline were reported. A marked reference range for hemoglobin 12.3-15.3 grams per deciliter (g/dL), lymphocytes absolute (Abs) 1.0-4.8 10^3/microliters (uL), neutrophils total, Abs, 1.8-8.5 10^3/uL, platelet 100-450 10^9/liter (L), total leukocyte 4.4-11 10^9/L.
Time Frame: From baseline up to 28 days after the last dose (up to approximately 24 weeks)
Population: Safety-evaluable population included all participants who received any amount of study treatment. Participants with at least 1 post-baseline assessment were included in the analysis. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Giredestrant + Palbociclib | Anastrozole + Palbociclib
Number analyzed (Participants) | 112 | 108
Participants
  Hemoglobin: Low: number analyzed (Participants) | 101 | 103
  Hemoglobin: Low | 3 | 1
  Hemoglobin: High: number analyzed (Participants) | 111 | 105
  Hemoglobin: High | 0 | 1
  Lymphocytes Abs: Low: number analyzed (Participants) | 95 | 91
  Lymphocytes Abs: Low | 9 | 2
  Lymphocytes Abs: High: number analyzed (Participants) | 90 | 88
  Lymphocytes Abs: High | 1 | 2
  Neutrophils, Total, Abs: Low: number analyzed (Participants) | 98 | 96
  Neutrophils, Total, Abs: Low | 43 | 38
  Platelet: Low | 0 | 0
  Total Leukocyte Count: Low | 15 | 11
  Total Leukocyte Count: High: number analyzed (Participants) | 104 | 105
  Total Leukocyte Count: High | 0 | 0

11. Secondary Outcome: Number of Participants With Shifts in Blood Chemistry Parameters From NCI-CTCAE Grade 0-2 at Baseline to Grade 3-4 at Post-baseline
Description: Blood chemistry parameters were measured per NCI CTCAE v5.0. Grade 0=normal, and Grades 1 to 4 represent worsening levels of parameter outside of normal range in the specified direction of abnormality (high & low are above & below the range, respectively). Number of participants with shift in blood chemistry values from grade 0-2 at baseline to grade 3-4 at post-baseline were reported. Marked reference range for albumin 32-45 grams per liter (g/L), alkaline phosphatase 20-130 units per liter (U/L), serum glutamic pyruvic transaminase (SGPT)/ alanine transaminase (ALT) 4-36 U/L, serum glutamic oxaloacetic transaminase (SGOT)/ aspartate transaminase (AST) 8-33 U/L, calcium 2.3-2.74 millimoles per liter (mmol/L), cholesterol 3.88-6.47mmol/L, creatinine 6-12 milligrams per liter (mg/L), glucose 3.9-6.1 mmol/L, potassium 3.5-5.0 mmol/L, sodium 135-147 mmol/L, bilirubin 2-21 micromoles per liter (μmol/L), triglycerides 0.11-2.15 mmol/L, & uric acid 2.7-7.3 milligrams per deciliter (mg/dL).
Time Frame: From baseline up to 28 days after the last dose (up to approximately 24 weeks)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Giredestrant + Palbociclib | Anastrozole + Palbociclib
Number analyzed (Participants) | 112 | 108
Participants
  Albumin: low: number analyzed (Participants) | 111 | 108
  Albumin: low | 1 | 0
  Alkaline Phosphatase: High | 0 | 0
  SGPT/ALT: High | 1 | 5
  SGOT/AST: High | 1 | 3
  Calcium: Low: number analyzed (Participants) | 102 | 101
  Calcium: Low | 0 | 3
  Calcium: High: number analyzed (Participants) | 109 | 103
  Calcium: High | 0 | 0
  Cholesterol: High: number analyzed (Participants) | 93 | 89
  Cholesterol: High | 0 | 0
  Creatinine: High | 0 | 1
  Glucose: Low | 0 | 0
  Potassium: Low: number analyzed (Participants) | 106 | 101
  Potassium: Low | 0 | 0
  Potassium: High: number analyzed (Participants) | 112 | 107
  Potassium: High | 0 | 0
  Sodium: Low: number analyzed (Participants) | 111 | 107
  Sodium: Low | 0 | 0
  Sodium: High: number analyzed (Participants) | 111 | 106
  Sodium: High | 0 | 0
  Bilirubin: High | 0 | 0
  Triglycerides: High: number analyzed (Participants) | 93 | 88
  Triglycerides: High | 1 | 0
  Uric Acid: High: number analyzed (Participants) | 87 | 86
  Uric Acid: High | 21 | 22

12. Secondary Outcome: Plasma Concentration of Giredestrant at Specified Timepoints
Time Frame: Window of Opportunity Phase: Day 1 (3 hours Postdose) and Day 15 (Predose) during Cycle 0 (the 15-day period in Window of Opportunity Phase is called Cycle 0 for PK analysis); Neoadjuvant Phase: Cycle 2 Day 1, Predose
Population: Pharmacokinetics (PK) evaluable population included all participants who received giredestrant and had at least one evaluable post-dose giredestrant plasma concentration. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliters (ng/mL)
Arm/Group | Giredestrant + Palbociclib
Number analyzed (Participants) | 108
nanograms per milliliters (ng/mL)
  Window of Opportunity Phase: Cycle 0 Day 1, 3-h Postdose | 81.8 (284)
  Window of Opportunity Phase: Cycle 0 Day 15, Predose: number analyzed (Participants) | 104
  Window of Opportunity Phase: Cycle 0 Day 15, Predose | 137 (61.1)
  Neoadjuvant Phase: Cycle 2 Day 1, Predose: number analyzed (Participants) | 99
  Neoadjuvant Phase: Cycle 2 Day 1, Predose | 130 (122)

ADVERSE EVENTS:
Time Frame: From baseline up to 28 days after the last dose (up to approximately 24 weeks)
Description: AEs are reported for the safety-evaluable population that was defined as all participants who received any amount of study treatment, grouped according to treatment received. All-cause mortality was also reported for the safety-evaluable population.
Arm/Group | Giredestrant + Palbociclib | Anastrozole + Palbociclib
All-Cause Mortality (participants affected / at risk) | 1/112 | 0/109
Serious Adverse Events (participants affected / at risk) | 5/112 | 2/109
Other Adverse Events (participants affected / at risk) | 99/112 | 93/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Giredestrant + Palbociclib (N=112) | Anastrozole + Palbociclib (N=109)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Uterine perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Giredestrant + Palbociclib (N=112) | Anastrozole + Palbociclib (N=109)
Anaemia (Blood and lymphatic system disorders) | 12 (13) | 6 (7)
Leukopenia (Blood and lymphatic system disorders) | 14 (20) | 16 (29)
Neutropenia (Blood and lymphatic system disorders) | 46 (77) | 44 (79)
Constipation (Gastrointestinal disorders) | 3 (3) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 8 (11) | 18 (25)
Nausea (Gastrointestinal disorders) | 16 (19) | 13 (15)
Vomiting (Gastrointestinal disorders) | 6 (6) | 1 (1)
Asthenia (General disorders) | 25 (28) | 27 (31)
Fatigue (General disorders) | 10 (10) | 18 (19)
Mucosal inflammation (General disorders) | 9 (9) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 6 (6)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 6 (6)
Alanine aminotransferase increased (Investigations) | 1 (1) | 9 (9)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 6 (6)
Neutrophil count decreased (Investigations) | 26 (39) | 24 (32)
White blood cell count decreased (Investigations) | 14 (19) | 10 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (13) | 21 (22)
Headache (Nervous system disorders) | 5 (5) | 9 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 6 (7) | 2 (2)
Hot flush (Vascular disorders) | 16 (16) | 16 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT04436744/Prot_SAP_001.pdf